CLINICAL TRIAL: NCT01231594
Title: A Rollover Study to Provide Continued Treatment With GSK2118436 to Subjects With BRAF Mutation-Positive Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114144
Record Dates: First submitted 2010-10-21; First posted 2010-11-01 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Cancer
Keywords: BRAF Inhibitor; Cancer; Safety; GSK2118436; BRAF mutation positive tumors
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Subjects who have received </= 8 weeks of GSK2118436 monotherapy in the parent study
  Interventions: Drug: GSK2118436
- Cohort B (Experimental): Subjects who have received >8 weeks of continuous treatment with GSK2118436 either as monotherapy or combination therapy with another approved anti-cancer agent
  Interventions: Drug: GSK2118436; Drug: Other approved anti-cancer agent
- Cohort C (Experimental): Subjects who have received >8 weeks of continuous treatment with GSK2118436 in combination with a MEK inhibitor, GSK1120212
  Interventions: Drug: GSK2118436; Drug: GSK1120212

INTERVENTIONS:
Drug: GSK2118436 — Study Drug
Drug: GSK1120212 — Study Drug
  Arms: Cohort C
Drug: Other approved anti-cancer agent — Study Drug
  Arms: Cohort B

SUMMARY:
This rollover study is designed to provide continued access to GSK2118436 for eligible subjects with BRAF mutation-positive tumors who have previously participated in a GlaxoSmithKline (GSK)-sponsored GSK2118436 study (parent study), who have no evidence of progressive disease and who have tolerated GSK2118436 in the parent study without significant toxicities. Subjects will be enrolled into the appropriate cohort based upon the treatment received in their parent study. Safety assessments (physical examinations, vital signs, 12-lead electrocardiograms, echocardiograms, clinical laboratory assessments, and monitoring of adverse events) will be made throughout the study. Clinical activity will be assessed using local standard of care imaging practices and the appropriate response criteria as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed written informed consent for this study
* Has demonstrated compliance with study drug(s), treatment visit schedules, and the requirements and restrictions listed in the consent form
* Is currently participating in a GSK-sponsored study of GSK2118436
* Currently has no evidence of progressive disease, as determined by the investigator, following previous treatment with GSK2118436 (either as monotherapy or as part of a combination treatment regimen)
* For Cohort C only: Subjects must have a calcium phosphate product (CPP) of <4.4 mmol^2/L^2 (55 mg^2/dL^2) if they are to continue treatment with GSK1120212
* Continued ability to swallow and retain orally administered study drug(s) and does not have any clinically significant GI abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Women of childbearing potential and men with reproductive potential must be willing to continue practicing acceptable methods of birth control during the study NOTE: Oral contraceptives are not reliable due to potential drug-drug interaction with GSK2118436
* Women of childbearing potential must have a negative serum pregnancy test at the time of transition to this study and before the first dose of study treatment
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Permanent discontinuation of GSK2118436 in the parent study due to toxicity or disease progression
* Local access to commercially available GSK2118436
* Currently receiving treatment with any prohibited medication(s)
* Any unresolved toxicity > Grade 2 (National Cancer Institute-Common Toxicity Criteria for Adverse Events [NCI-CTCAE], version 4.0) from parent study treatment, except for alopecia, will need to be approved by the GSK Medical Monitor
* Uncontrolled diabetes, hypertension or other medical conditions at the time of transition to this study that may interfere with assessment of toxicity
* Presence of rheumatoid arthritis
* Corrected QT (QTc) interval >/= 480 msec at the time of transition to this study
* Left ventricular ejection fraction (LVEF) </= institutional lower limit of normal (LLN) by ECHO at the time of transition to this study
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system at the time of transition to this study
* Pregnant or lactating female
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions at the time of transition to this study that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator or GSK Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2010-11-05 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, as a measure of safety and tolerability | From date of transition into this Rollover study until 28 days following the last dose. Subjects may continue to receive study medication until disease progression, death or unacceptable adverse event; there is no time limit for this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (41):
- United States (22):
  - Novartis Investigative Site, Goodyear, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Tacoma, Washington
- Australia (6):
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Lille, France
- Germany (3):
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
- Novartis Investigative Site, Napoli, Campania, Italy
- Poland (2):
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Warsaw
- Spain (3):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
- United Kingdom (2):
  - Novartis Investigative Site, Headington
  - Novartis Investigative Site, London